CLINICAL TRIAL: NCT05136391
Title: A Phase I Study to Evaluate the Safety, Biodistribution, Radiation Dosimetry, and Pharmacokinetics of XTR003 in Healthy Chinese Volunteers
Brief Title: A Phase I Study to Evaluate XTR003 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STB-XTR003-101
Record Dates: First submitted 2021-11-23; First posted 2021-11-29 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: coronary artery disease; positron emission tomography (PET)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XTR003 (Experimental): Administration and investigation of myocardial fatty acid radiotracer
  Interventions: Drug: XTR003

INTERVENTIONS:
Drug: XTR003 — Single dose of 8.0-10 mCi of XTR003 will be injected on the first day of the study (Day 1). Serial whole-body PET imaging will be acquired after dose injection.

SUMMARY:
18F-FDG PET imaging is now considered the most effective method used in the clinical evaluation of viable myocardium. However, the need for fasting or glucose and insulin loading in the 18F-FDG PET protocol makes it unfavorable for a certain group of patients (i.e., insulin-resistance and diabetic patients). XTR003 is a fatty acid analog used for PET imaging, developed at the Beijing Anzhen Hospital affiliated to Sinotau Pharmaceutical Group. XTR003 is a promising fatty acid analog and perhaps have a potential clinical utility in the evaluation of viable myocardium. This phase I study investigated the safety, biodistribution, radiation dosimetry and Pharmacokinetics of XTR003 in 10 Chinese normal healthy volunteers both male and female between the ages of 18-40.

DETAILED DESCRIPTION:
XTR003 is a PET imaging radiopharmaceutical agent used to trace myocardial fatty acid metabolism. XTR003 is a modified fatty acid that enters the myocytes and passes through mitochondrial membrane by the same process as the natural existing fatty acids and then undergoes partial β-oxidation before being trapped in the mitochondria. In preclinical study XTR003 showed high myocardial uptake and retention [1].

This is a phase I study, the study will be open-label, nonrandomised, single-arm, single-center clinical study. Subjects will receive single dose of XTR003.

Safety, biodistribution, radiation dosimetry and Pharmacokinetics was investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 18-40 years
2. Normal electrocardiogram and echocardiography
3. Normal vital signs and physical examination
4. No any major illness
5. No clinically significant abnormalities in laboratory tests
6. No clinically significant anomalies in 12-lead ECG
7. Females of child bearing possibility should adopt effective medically approved contraceptive methods to prevent pregnancy for at least 6 months before the study and after the study
8. Voluntarily signed written consent from all subjects

Exclusion Criteria:

1. Pregnancy or lactating woman
2. History of cardiovascular disease
3. History of any brain disease
4. History of coagulopathy
5. History of liver or gastrointestinal diseases or other factors that can interfere with drug absorption, distribution, excretion or metabolism
6. Past history of cancer
7. History of drug allergy
8. History of drug abuse or alcohol dependance
9. Any medications and treatments that may interfere with the test data or may cause serious side effects
10. Human immunodeficiency virus (HIV), hepatitis C or syphilis antibody test positive, hepatitis B surface antigen positive
11. Exposure to significant occupational radiation (e.g >50 mvs/year) or exposure radioactive substances for therapeutic or research purposes over the past 10 years
12. Use of health products or medications (eg. coenzyme Q10, etc.) that have an effect on myocardial energy metabolism within 1 week
13. Hospital admission due to illness during the screening period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of healthy Chinese adults after a single dose of XTR003 intravenous injection. On Day1 of the study all subjects received a single dose 8.0-10 mCi of XTR003 intravenously. | 0 to 14 days post injection
  All subjects returned to the hospital on Day 2 and Day 7 after XTR003 injection for safety observation that included: Physical examination, vital signs monitoring, blood troponin-I levels, routine blood test, blood biochemistry test, routine urine test, and 12-lead electrocardiogram. On Day 14 all subjects were telephoned for the final follow-up. All adverse events after enrolment in the study will be documented.

SECONDARY OUTCOMES:
To investigate the biodistribution of XTR003 | 0 to 5 hours
  XTR003 biodistribution will be determined by whole body PET imaging acquisition at point time intervals at 0-60, 120, 150, 240, and 270 minutes. Venous blood collection of 10 ml from each subject at set time points at 1.5, 3, 5, 10, 30, 60, and 120 minutes after administration and at 4 and 7 hours for radioactivity measurement. Urine collection will begin immediately after injection up to ~ 7.25 hours for radioactivity measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Shoup TM, Elmaleh DR, Bonab AA, Fischman AJ. Evaluation of trans-9-18F-fluoro-3,4-Methyleneheptadecanoic acid as a PET tracer for myocardial fatty acid imaging. J Nucl Med. 2005 Feb;46(2):297-304. PMID 15695790
- [Derived] Mou T, Meng J, Lin C, Xie X, Hsu B, Zhang X. XTR003, a fatty acid metabolism PET tracer: A phase I study to evaluate the safety, biodistribution, radiation dosimetry, and pharmacokinetics in healthy volunteers. J Nucl Cardiol. 2025 Apr;46:102144. doi: 10.1016/j.nuclcard.2025.102144. Epub 2025 Feb 7. PMID 39923833